CLINICAL TRIAL: NCT02484261
Title: Pilot Study to Evaluate the Tolerability of Velcade (Bortezomib) and Pravastatin for the Treatment of Relapsed Leukemia Following Allogeneic Hematopoietic Stem Cell Transplantation in Children
Brief Title: Monitoring and Treatment of Relapsed Leukemia Following Allogeneic Hematopoietic Stem Cell Transplantation in Children
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Contractual/Funding/Accrual
Sponsor: Reuven Schore (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry); Hyundai Hope On Wheels (Other)
Responsible Party: Sponsor-Investigator, Reuven Schore, MD, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Pro00004062
Record Dates: First submitted 2015-06-24; First posted 2015-06-29 (Estimated); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Leukemia
Keywords: childhood leukemia; relapsed leukemia; Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Leukemia | interventions — Bortezomib; Pravastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Monitoring phase (No Intervention): Patients who have received a Stem cell transplant for Hematologic malignancies will be monitored for signs of relapse with blood tests for CD34+ chimerism. Patients with signs of relapse will have bone marrow aspirate and/or other appropriate tests to confirm presence of relapse. All patients who are confirmed to have relapsed and meet eligibility criteria to receive study drug will be eligible to receive treatment on the treatment arm.
- Treatment phase (Experimental): Patients with confirmed disease will initiate therapy with bortezomib and pravastatin, a regimen that has efficacy in treatment of leukemia and graft-versus-host disease, while sparing healthy donor hematopoietic stem cells may improve the dismal survival of relapse post allogeneic transplant. Depending on response, patients may receive up to 13 cycles of therapy
  Interventions: Drug: Bortezomib; Drug: Pravastatin

INTERVENTIONS:
Drug: Bortezomib — 1.3 mg/m2/dose subcutaneously (SQ) daily (total 4 doses) on Days 1, 4, 8 and 11 (+/- 1 day with at least 72 hours between doses) q3 weeks. (For patients continuing to receive drug in cycles 6 or greater, at investigator discretion, the schedule may be changed to 1.3 mg/m2/dose SQ daily (total 3 doses) on Days 1, 8, and 15 (+/- 1 day with at least 72 hours between doses) every 4 weeks in an effort to decrease risk of peripheral neuropathy.)
  Other Names: Velcade
  Arms: Treatment phase
Drug: Pravastatin — 10 mg for age < 8 years, 20 mg for age 8-<13 years, 40 mg for ages >14 years
  Arms: Treatment phase

SUMMARY:
This study aims to monitor patients for relapse of the leukemia following allogeneic Hematopoietic Stem Cell Transplantation (HSCT) in order to identify patients early in relapse, with a low burden of disease, when interventions may be more successful by monitoring of peripheral blood lineage specific chimerism. Once disease has been confirmed, patients will initiate a novel combination of bortezomib and pravastatin.

DETAILED DESCRIPTION:
Patients will be enrolled on this study at the time of transplantation. Following HSCT, CD34+ chimerism in peripheral blood will be monitored in real time at scheduled intervals. If chimerism of CD34+ cells diminishes post-HSCT or clinical signs or symptoms of relapsed leukemia, relapse in bone marrow will be confirmed, after which immunosuppression will be withdrawn and treatment initiated with bortezomib and pravastatin. Patients will be monitored for disease response until 1 year post-HSCT or post-study therapy. Patients with confirmed relapse post-HSCT will also be eligible to enroll and receive novel combination.

ELIGIBILITY:
Inclusion Criteria to enter study:

* Voluntary written informed consent by patient or legal guardian (as appropriate) before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
* Female patients who:

  * Are postmenopausal for at least 1 year before the Screening visit, OR
  * Are surgically sterile, OR
  * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 30 days after the last dose of study treatment, OR agree to completely abstain from heterosexual intercourse

OR Male patients, even if surgically sterilized (i.e., status postvasectomy), who:

* Agree to practice effective barrier contraception during the entire study treatment period and through 30 days after the last dose of study treatment, OR
* Agree to completely abstain from heterosexual intercourse

  * Lansky(if age <15)/Karnofsky (if age >16 yr) performance status > 50%
  * Hepatic function: total bilirubin ≤ 2.5 mg/dl, and ALT/AST < or equal to 5 x the upper limit of normal
  * Renal function: Creatinine clearance > 60 ml/min/1.73 m2 (as determined by 24 hour collection or nuclear (glomerular filtration rate) GFR or Cystatin C calculation)
  * Cardiac function: LVEF > 50% or LVSF > 27%
  * Pulmonary function tests: DLCO and FEV1 > 50% (if able to perform PFTs, if not able to perform PFTs SAO2> 94% on room air).
  * Acute leukemia or Myelodysplastic syndrome (MDS)

Inclusion Criteria to initiate therapy with bortezomib and pravastatin

* Lansky performance status (if age < 15) /Karnofsky (if age >16 yr) performance status > 50%
* Hepatic function: total bilirubin ≤ 2.5 mg/dl, and ALT/AST < or equal to 5 x the upper limit of normal (ULN)
* Renal function: Cr < ULN for age
* Relapse of systemic disease documented by any of the following: morphology, flow cytometry, cytogenetics and/or FISH.
* Patient has a platelet count of more than 20,000/μL within 7 days before enrollment. Patients may be transfused prior to this evaluation but may not be platelet refractory at enrollment.
* Patient has an absolute neutrophil count of greater than 500 /μL within 7 days before enrollment.
* Patients with confirmed relapse post-HSCT who were not previously enrolled on monitoring portion of protocol, will also be eligible to enroll and receive novel combination if entry criteria met at time of relapse.

Exclusion Criteria:

Patients meeting any of the following exclusion criteria are not to be treated on the study:

* Patient has greater than or equal to Grade 2 peripheral neuropathy
* Patient had myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening must be documented by the investigator as not medically relevant.
* Patient has hypersensitivity to bortezomib, boron, or mannitol.
* Female patients who are lactating or pregnant.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Evidence of residual or relapse of another malignancy(other than the hematological malignancy which is the indication for stem cell transplant)at the time of transplant preparative regimen initiation
* Participation in clinical trials with other investigational agents not included in this trial, within 14 days of the start of bortezomib/pravastatin and throughout the duration of therapy.
* Radiation therapy within 3 weeks before start of bortezomib/pravastatin. Enrollment of subjects who require concurrent radiotherapy (which must be localized in its field size) should be deferred until the radiotherapy is completed and 3 weeks have elapsed since the last date of therapy.

Ages: 22 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2015-05; Primary Completion 2018-05-18 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 3 years
  Tolerability of bortezomib and pravastatin in pediatric relapsed leukemia patients following allogeneic transplantation

SECONDARY OUTCOMES:
Number of relapses that are detected by CD34+ chimerism before clinical symptoms | 3 years
  The sensitivity of detection of recurrent acute leukemia in pediatric patients by peripheral blood CD34+ chimerism in pediatric patients following allogeneic HSCT

OTHER OUTCOMES:
The number of patients who respond to bortezomib and pravastatin treatment for relapsed acute leukemia as defined by those that achieve complete response, partial response or stable disease | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Reuven Schore, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States